CLINICAL TRIAL: NCT04098835
Title: A Pilot Study of a Strategy and Computer-based Intervention to Enhance Daily Cognitive Functioning After Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-06020310
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASCEND (Experimental): ASCEND combines computer-based cognitive training exercises, homework exercises to enhance cognition, and coaching sessions delivered in-person and via telephone/videoconference by a neuropsychologist. ASCEND includes 24 total computer training sessions of 30 minutes each, for a total of 12 hours. ASCEND includes 8 coaching sessions of 45 minutes each. The computer exercises aim to improve attention, working memory (WM), and cognitive control through a series of engaging and interactive computer games (e.g., card games, driving simulation). The homework exercises and coaching sessions aim to assist the participant in generalizing and transferring skills from the computer exercises to daily life and to develop further strategies to compensate for attention and WM difficulties in daily life.
  Interventions: Behavioral: ASCEND

INTERVENTIONS:
Behavioral: ASCEND — ASCEND is a behavioral intervention that combines computer-based cognitive exercise, strategy coaching with a neuropsychologist, and homework exercises in order to improve attention, working memory, and cognitive control after stroke.

SUMMARY:
This is an initial pilot study to test feasibility, participant engagement and satisfaction, and clinical and neurobiological target engagement of a behavioral treatment called "ASCEND" that combines computer-based cognitive training and coaching of cognitive strategies to improve daily cognitive functioning in individuals with stroke.

ELIGIBILITY:
Inclusion Criteria:

* History of first-time stroke, minimum of 6 months prior to enrollment
* English speaking
* Ability to comprehend sufficiently to participate in the treatment.
* Subjective or objective evidence of mild cognitive impairment
* Willingness to participate in full study duration
* Has computer that meets specification for the training program software.
* Physically able to operate a computer keyboard and mouse.
* Not concurrently receiving other cognitive rehabilitation services
* Cognitively able to perform basic self-care activities (e.g., dressing, grooming, eating).

Exclusion Criteria:

* History of neurologic disease other than stroke
* History of severe mental illness or substance use disorder, or current major depressive episode.
* History of dementia or dependence in basic self-care activities due to cognitive deficits
* Contraindications to MRI

Ages: 45 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Participant satisfaction with ASCEND, as measured by the Client Satisfaction Questionnaire-8 (CSQ-8) | 5 weeks (at the conclusion of treatment)
  The CSQ-8 is a self-report measure of participant satisfaction with the intervention. Scores range from 8-32 with higher scores indicating greater satisfaction.
Participant impression of ASCEND as a credible treatment to improve cognition, as measured by the Credibility and Expectancy Questionnaire (CEQ). | 5 weeks (at the conclusion of treatment)
  The CEQ is a self-report measure that assesses participants' perceived benefit and improvement from the intervention. Each item is scored on a 1-9 Likert-type scale or as a percentage rating from 0% to 100% in 10% increments.

SECONDARY OUTCOMES:
Change in auditory attention and working memory, as measured by the Digit Span test | Baseline, 5 weeks
  Performance-based measure of attention/working memory with scores ranging from 0-48, with higher scores indicating better performance.
Change in visual attention and working memory, as measured by the Symbol Span test | Baseline, 5 weeks
  Performance-based measure of attention/working memory with scores ranging from 0-50, with higher scores indicating better performance.
Change in divided attention and working memory, as measured by the Symbol-Digit Modalities Test | Baseline, 5 weeks
  Performance-based measure of divided attention/working memory with scores ranging from 0-120, with higher scores indicating better performance.
Change in divided attention and processing speed, as measured by the Trail Making Test | Baseline, 5 weeks
  Performance-based and timed measure of divided attention/processing speed with lower scores indicating better performance (faster completion time).
Change in selective attention and inhibitory control, as measured by the Stroop Test | Baseline, 5 weeks
  Performance-based and timed measure of selective attention and inhibition, with higher scores indicating better performance.
Change in rapid working memory and mental arithmetic, as measured by the Paced Auditory Serial Addition Test (PASAT) | Baseline, 5 weeks
  Performance-based and timed measure of rapid working memory, with higher scores indicating better performance.
Change in attention and working memory as measured by the Mental Control test | Baseline, 5 weeks
  Performance-based measure of simple auditory attention and working memory. Scores range from 0-12 with higher scores indicating better performance.
Change in executive functioning as measured by the Weekly Calendar Planning Activity | Baseline, 5 weeks
  Performance-based measure of executive functioning. Higher scores indicate better performance.
Change in self-reported executive functioning as measured by the Behavior Rating Inventory of Executive Function-Adult | Baseline, 5 weeks
  Self-report measure of executive functioning. Higher scores indicate greater problems with executive dysfunction in daily life.
Change in self-reported cognitive symptoms due to stroke, as measured by the Patient Reported Evaluation of Cognitive State (PRECIS). | Baseline, 5 weeks
  Self-report measure of cognitive difficulties after stroke. Scores range from 0-128 with higher scores indicating greater cognitive problems in daily life due to stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Jaywant, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- NewYork-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No